CLINICAL TRIAL: NCT03637465
Title: A Randomized Trial of a Comprehensive Multi-level Intervention to Increase Water Access and Appeal in Community Recreation Centers
Brief Title: Increasing Water Access and Appeal in Community Recreation Centers
Acronym: Hydrate Philly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia Department of Public Health (Other Government)
Collaborators: Stanford University (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Hannah Lawman, Director of Research and Evaluation, Get Healthy Philly, Philadelphia Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 49200; 74395 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2018-07-31; First posted 2018-08-20 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Health Behavior
Keywords: hydration; water intake; sugar sweetened beverages; youth; children
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This cluster RCT involves 14 matched pairs; study recruitment and randomization occurs at the recreation center-level. Participating sites are matched based on center size, summer program enrollment, presence of indoor gym, neighborhood income & race/ethnicity. Then, an intervention site and control site are randomly determined by a coin flip within each pair.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrate Philly Intervention (Experimental): Intervention group that receives hydration station intervention
  Interventions: Behavioral: Hydrate Philly
- Control (No Intervention): Control group that receives no intervention, but observational data is collected; converted to wait-listed intervention status after enrollment and randomization was completed

INTERVENTIONS:
Behavioral: Hydrate Philly — Hydrate Philly is a multi-component intervention that includes water safety testing, provision of 1-2 hydration stations per recreation center, distribution of reusable water bottles for youth, a campaign to promote the acceptability of tap water, and the reduction of access to competing unhealthy beverages through vending machine standards and discouraging "black bags" (characteristic small, black, plastic bags provided to customers with their corner store purchases, typically including a sugar sweetened beverage and/or unhealthy snack foods).
  Arms: Hydrate Philly Intervention

SUMMARY:
This study is a cluster randomized controlled trial with n=28 City of Philadelphia recreation centers (14 matched pairs) designed to determine the effectiveness of a comprehensive multi-level intervention to increase water access and appeal in community recreation centers on 1) center-level water intake as measured by water meters, and 2) purchase of outside beverages as measured by observations of recreation center youth.

ELIGIBILITY:
Inclusion Criteria:

* Recreation center is located in a low-income neighborhood in the City of Philadelphia, defined by ≥20% of the residents in the zip code at or below Federal Poverty Level
* Recreation center includes both summer and after-school programming
* Recreation center is willing to comply with City of Philadelphia Healthy Vending standards and discourage sugar sweetened beverage consumption
* Recreation center has water lines appropriate for installing indoor hydration stations

Exclusion Criteria:

* Unwilling to accept randomization

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Center water consumption | Three measurement periods, each lasting 2 weeks, will occur: baseline (2-4 months pre-intervention), mid-point (3-5 months post intervention), and post (7-10 months post intervention).
  Change in average gallons of water per day used at the center drinking water source as measured by flow meters over each 2-week measurement period.
Outside beverages during programs | Three measurement periods, each lasting 2 weeks, will occur: baseline (2-4 months pre-intervention), mid-point (3-5 months post intervention), and post (7-10 months post intervention).
  Changes in the average number of sugary beverages per day brought to summer camp.

SECONDARY OUTCOMES:
Single use beverage containers | Three measurement periods, each lasting 2 weeks, will occur: baseline (2-4 months pre-intervention), mid-point (3-5 months post intervention), and post (7-10 months post intervention).
  Average number of single use containers (bottled water + sugary beverages) as measured by recreation center staff daily reports
Staff consumption of sugary beverages | Three measurement periods, each lasting 2 weeks, will occur: baseline (2-4 months pre-intervention), mid-point (3-5 months post intervention), and post (7-10 months post intervention).
  Change in frequency of staff consumption of sugary beverages (i.e., number of days in past 30 days with sugary beverages consumed) as measured by the Beverage Intake Questionnaire (BEVQ-15) survey assessing past 30 day recall of overall beverage intake. Range is 0 - 30 with higher values indicating more days sugary beverages were consumed.
Fountain related maintenance problems | Questionnaire administered 2-5 times per site up to 8 months post intervention
  Average maintenance rating of scale with 8 items (4-point scale; i.e., everyday, 3-4 times, once or twice, or never) at post as measured by staff self-report. Subscales include average routine maintenance (3 items) versus average maintenance problems (5 items).
Center attendance | Three measurement periods, each lasting 2 weeks, will occur: baseline (2-4 months pre-intervention), mid-point (3-5 months post intervention), and post (7-10 months post intervention).
  The number of youth attending the recreation center program daily

CONTACTS AND LOCATIONS:
Overall Officials: Hannah G Lawman, PhD, Principal Investigator — Philadelphia Department of Public Health, Division of Chronic Disease Prevention
Locations (1):
- Philadelphia Department of Public Health, Division of Chronic Disease Prevention, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawman HG, Grossman S, Lofton X, Tasian G, Patel AI. Hydrate Philly: An Intervention to Increase Water Access and Appeal in Recreation Centers. Prev Chronic Dis. 2020 Feb 20;17:E15. doi: 10.5888/pcd17.190277. PMID 32078503
- [Derived] Lawman HG, Lofton X, Grossman S, Root M, Perez M, Tasian G, Patel A. A randomized trial of a multi-level intervention to increase water access and appeal in community recreation centers. Contemp Clin Trials. 2019 Apr;79:14-20. doi: 10.1016/j.cct.2019.02.003. Epub 2019 Feb 13. PMID 30771559

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT03637465/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03637465/SAP_001.pdf